CLINICAL TRIAL: NCT00619359
Title: A Phase III, Randomized, Double-Blind, Active-Controlled, Parallel-Group Study, Conducted Under In-House Blinding Conditions, to Examine the Safety, Tolerability, and Efficacy of a Single Dose of Intravenous MK-0517 for the Prevention of Chemotherapy-Induced Nausea and Vomiting (CINV) Associated With Cisplatin Chemotherapy
Brief Title: Evaluation of Fosaprepitant (MK0517) in Single Dose Schedule (0517-017)
Acronym: EASE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0517-017; MK0517-017; 2007_594
Record Dates: First submitted 2008-01-28; First posted 2008-02-21 (Estimated); Results first posted 2010-02-12 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting (CINV)
MeSH Terms: conditions — Vomiting | interventions — Dexamethasone; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Arm 1: study medication
  Interventions: Drug: Comparator: fosaprepitant dimeglumine; Drug: Dexamethasone; Drug: Ondansetron
- 2 (Active Comparator): Arm 2: Active comparator
  Interventions: Drug: Comparator: Aprepitant; Drug: Dexamethasone; Drug: Ondansetron

INTERVENTIONS:
Drug: Comparator: fosaprepitant dimeglumine — single IV dose of 150 mg of fosaprepitant dimeglumine on Day 1.
  Arms: 1
Drug: Comparator: Aprepitant — Aprepitant 3-day dosing oral regimen (125 mg on Day 1 followed by 80 mg on Days 2 and 3).
  Arms: 2
Drug: Dexamethasone — Oral dose of 12 mg of dexamethasone on Day 1, 8 mg on Day 2, and 8 mg twice a day on Days 3-4.
  Arms: 1
Drug: Dexamethasone — Oral dose of 12 mg of dexamethasone on Day 1, and 8 mg on Days 2-4.
  Arms: 2
Drug: Ondansetron — single IV dose of 32 mg of ondansetron on Day 1.

SUMMARY:
The purpose of this study is to examine the safety, tolerability, and efficacy of MK0517 to prevent Chemotherapy-Induced Nausea and Vomiting (CINV) associated with Cisplatin chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female and is at least 18 years of age; scheduled to receive his or her first course of cisplatin chemotherapy at a dose of 70 mg/m2 or higher; predicted life expectancy of 3 months or greater
* Patient is post menopausal or, if premenopausal, must use double-barrier contraception

Exclusion Criteria:

* Patient has symptomatic primary or metastatic CNS malignancy
* Patient has received or will receive Radiation therapy to the abdomen or pelvis in the week prior to Treatment Day 1 though Day 6
* Patient has vomited in the 24 hours prior to treatment Day 1
* Patient has an active infection; Patient uses illicit drugs or has current evidence of alcohol abuse
* Patient is pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2322 (Actual)
Dates: Start 2008-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Grunberg S, Chua D, Maru A, Dinis J, DeVandry S, Boice JA, Hardwick JS, Beckford E, Taylor A, Carides A, Roila F, Herrstedt J. Single-dose fosaprepitant for the prevention of chemotherapy-induced nausea and vomiting associated with cisplatin therapy: randomized, double-blind study protocol--EASE. J Clin Oncol. 2011 Apr 10;29(11):1495-501. doi: 10.1200/JCO.2010.31.7859. Epub 2011 Mar 7. PMID 21383291

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 149 medical centers worldwide. The recruitment period was from 12 Feb 08 through 8 Jun 09.
Pre-assignment Details: Cisplatin-naïve patients scheduled to receive cisplatin chemotherapy at a dose of 70 mg/m2 or higher for a documented solid malignancy were screened up to 30 days prior to initiation of chemotherapy. Screening included a complete medical history and physical exam. Informed consent was obtained for patients who agreed to participate in the study.
Groups:
- Fosaprepitant: Fosaprepitant dimeglumine 150 mg IV, ondansetron 32 mg IV, and dexamethasone 12 mg by mouth (PO) on Day 1, dexamethasone 8 mg PO on Day 2, and dexamethasone 16 mg PO on Days 3 and 4.
- Aprepitant: Aprepitant 125 mg by mouth (PO), ondansetron 32 mg IV, and dexamethasone 12 mg PO on Day 1, aprepitant 80 mg PO and dexamethasone 8 mg PO on Days 2 and 3, dexamethasone 8 mg PO on Day 4.
Period: Overall Study
Arm/Group | Fosaprepitant | Aprepitant
Started | 1147 | 1175
Completed | 1080 | 1094
Not Completed | 67 | 81
Not completed — Adverse Event | 32 | 36
Not completed — Lost to Follow-up | 12 | 16
Not completed — Physician Decision | 0 | 7
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 19 | 20
Not completed — Progressive Disease | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fosaprepitant | Aprepitant | Total
Number analyzed (Participants) | 1147 | 1175 | 2322
Age, Continuous [Mean (Full Range); unit: years] | 55.2 [19 to 86] | 55.9 [19 to 82] | 55.6 [19 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 425 | 427 | 852
  Male | 722 | 748 | 1470
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 32 | 33 | 65
  Asian | 296 | 306 | 602
  Black or African American | 21 | 22 | 43
  Multi-Racial | 149 | 157 | 306
  Native Hawaiian or Pacific Islander | 1 | 2 | 3
  White | 648 | 655 | 1303
History of Motion Sickness [Number; unit: Participants] — Includes treated patients only.
  Participants
    Yes | 0 | 3 | 3
    No | 1143 | 1166 | 2309
    No Data - Assessment Not Completed | 4 | 6 | 10
History of Vomiting with Pregnancy [Number; unit: Participants] — Measure is specific to female treated patients only.
  Participants
    Yes | 3 | 3 | 6
    No | 420 | 421 | 841
    Female Patients with No Data - No Assessment | 2 | 3 | 5
    Not Applicable - Male Patients | 722 | 748 | 1470

OUTCOME MEASURES:

1. Primary Outcome: A Complete Response (no Vomiting and no Use of Rescue Therapy) Overall (in the 120 Hours Following Initiation of Cisplatin).
Description: The number of patients who reported No Vomiting and No Use of Rescue Therapy in the 120 hours following initiation of cisplatin chemotherapy.
Time Frame: Overall (in the 120 hours following initiation of cisplatin chemotherapy).
Population: FAS (Full Analysis Set) patient population was used for all efficacy evaluations and included patients who: 1) received at least one dose of study therapy, 2) received cisplatin chemotherapy, and 3) had at least one post-treatment efficacy assessment.
Measure: Number; unit: Participants
Arm/Group | Fosaprepitant | Aprepitant
Number analyzed (Participants) | 1106 | 1134
Participants | 795 | 820
Statistical Analysis 1: Comparison: Fosaprepitant vs Aprepitant; Test type: Non-Inferiority or Equivalence — If the CI for the difference in response rates (Fosaprepitant minus Aprepitant), calculated using the methodology of Miettinen and Nurminen, had a lower limit ≥7 percentage points, fosaprepitant was considered at least as effective as aprepitant for Complete Response in the overall phase. Study had 90% power to detect non-inferiority for this outcome measure; Risk Difference (RD) = -0.4, 95% CI [-4.1 to 3.3], Standard Error of Mean 3.7

2. Secondary Outcome: A Complete Response (no Vomiting and no Use of Rescue Therapy) in the Delayed Phase (25 to 120 Hours Following Initiation of Cisplatin).
Description: The number of patients who reported No Vomiting and No Use of Rescue Therapy in the 25 to 120 hours following initiation of cisplatin chemotherapy.
Time Frame: Delayed phase (25 to 120 hours following initiation of cisplatin).
Population: FAS (Full Analysis Set) patient population was used for all efficacy evaluations and included patients who: 1) received at least one dose of study therapy, 2) received cisplatin chemotherapy, and 3) had at least one post-treatment efficacy assessment. 1 patient (aprepitant group) had no delayed phase data, and was not included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Fosaprepitant | Aprepitant
Number analyzed (Participants) | 1106 | 1133
Participants | 822 | 841
Statistical Analysis 1: Comparison: Fosaprepitant vs Aprepitant; Test type: Non-Inferiority or Equivalence — If the CI for the difference in response rates, calculated using the methodology of Miettinen and Nurminen, had a lower limit ≥7.3 percentage points, fosaprepitant was considered at least as effective as aprepitant for Complete Response in the delayed phase; Risk Difference (RD) = 0.1, 95% CI [-3.5 to 3.7], Standard Error of Mean 3.6

3. Secondary Outcome: No Vomiting Overall (in the 120 Hours Following Initiation of Cisplatin)
Description: The number of patients who reported No Vomiting in the 120 hours following initiation of cisplatin chemotherapy.
Time Frame: Overall (the 120 hours following initiation of cisplatin chemotherapy)
Population: FAS (Full Analysis Set) patient population was used for all efficacy evaluations and included patients who: 1) received at least one dose of study therapy, 2) received cisplatin chemotherapy, and 3) had at least one post-treatment efficacy assessment. 2 patients (aprepitant group) had no vomiting data, and were excluded from this analysis.
Measure: Number; unit: Participants
Arm/Group | Fosaprepitant | Aprepitant
Number analyzed (Participants) | 1106 | 1132
Participants | 806 | 844
Statistical Analysis 1: Comparison: Fosaprepitant vs Aprepitant; Test type: Non-Inferiority or Equivalence — If the CI for the difference in response rates, calculated using the methodology of Miettinen and Nurminen, had a lower limit ≥8.2 percentage points, fosaprepitant was considered at least as effective as aprepitant for No Vomiting in the overall phase; Risk Difference (RD) = -1.7, 95% CI [-5.3 to 2.0], Standard Error of Mean 3.6

ADVERSE EVENTS:
Time Frame: AEs were collected starting from the Pre-Study Visit (Day -30 to Day -1) up to 14 days after the patient's last dose of study drug.
Description: Severe infusion site pain, severe infusion site erythema and/or severe infusion site induration, as well as any episode of infusion site thrombophlebitis were designated Events of Clinical Interest (ECI) and evaluated using a predefined severity assessment scale.
Groups:
- Fosaprepitant: Fosaprepitant dimeglumine 150 mg IV, ondansetron 32 mg IV, and dexamethasone 12 mg by mouth (PO) on Day 1, dexamethasone 8 mg PO on Day 2, and dexamethasone 16 mg PO on Days 3 and 4.
  4 patients from the fosaprepitant regimen were randomized to the study, but discontinued before receiving study drug. These patients were excluded from the Adverse Event tables.
- Aprepitant: Aprepitant 125 mg by mouth (PO), ondansetron 32 mg IV, and dexamethasone 12 mg PO on Day 1, aprepitant 80 mg PO and dexamethasone 8 mg PO on Days 2 and 3, dexamethasone 8 mg PO on Day 4.
  6 patients from the aprepitant regimen were randomized to the study, but discontinued before receiving study drug. These patients were excluded from the Adverse Event tables.
Arm/Group | Fosaprepitant | Aprepitant
Serious Adverse Events (participants affected / at risk) | 148/1143 | 157/1169
Other Adverse Events (participants affected / at risk) | 636/1143 | 679/1169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fosaprepitant (N=1143) | Aprepitant (N=1169)
Anaemia (Blood and lymphatic system disorders) | 3 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 18 | 27
Leukopenia (Blood and lymphatic system disorders) | 4 | 2
Neutropenia (Blood and lymphatic system disorders) | 17 | 13
Pancytopenia (Blood and lymphatic system disorders) | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 8
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 3
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Regurgitation (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 13 | 7
Asthenia (General disorders) | 4 | 8
Chest pain (General disorders) | 1 | 1
Death (General disorders) | 2 | 5
Fatigue (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 3 | 2
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 1 | 2
Pyrexia (General disorders) | 1 | 2
Suprapubic pain (General disorders) | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 2
Diarrhoea infectious (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 5
Gastroenteritis shigella (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Incision site abscess (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Perineal abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 9
Postoperative wound infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 5 | 1
Septic shock (Infections and infestations) | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Wound infection (Infections and infestations) | 0 | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 2 | 1
Blood potassium decreased (Investigations) | 0 | 2
Haemoglobin decreased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 3 | 5
Dehydration (Metabolism and nutrition disorders) | 12 | 9
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 2
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 2
Cognitive disorder (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 2 | 1
Dizziness (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 3 | 2
Renal failure acute (Renal and urinary disorders) | 3 | 1
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 0 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Arterial occlusive disease (Vascular disorders) | 1 | 0
Arterial thrombosis (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0
Flushing (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 2
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 3
Peripheral embolism (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fosaprepitant (N=1143) | Aprepitant (N=1169)
Anaemia (Blood and lymphatic system disorders) | 17 | 7
Leukopenia (Blood and lymphatic system disorders) | 14 | 16
Neutropenia (Blood and lymphatic system disorders) | 28 | 25
Thrombocytopenia (Blood and lymphatic system disorders) | 17 | 14
Tinnitus (Ear and labyrinth disorders) | 19 | 10
Abdominal pain (Gastrointestinal disorders) | 34 | 35
Abdominal pain upper (Gastrointestinal disorders) | 46 | 29
Constipation (Gastrointestinal disorders) | 119 | 111
Diarrhoea (Gastrointestinal disorders) | 86 | 95
Dyspepsia (Gastrointestinal disorders) | 50 | 38
Gastritis (Gastrointestinal disorders) | 12 | 9
Nausea (Gastrointestinal disorders) | 64 | 78
Stomatitis (Gastrointestinal disorders) | 20 | 18
Vomiting (Gastrointestinal disorders) | 62 | 58
Asthenia (General disorders) | 94 | 129
Chest pain (General disorders) | 15 | 18
Fatigue (General disorders) | 53 | 56
Infusion site pain (General disorders) | 16 | 1
Mucosal inflammation (General disorders) | 22 | 32
Pain (General disorders) | 11 | 10
Pyrexia (General disorders) | 22 | 23
Accidental overdose (Injury, poisoning and procedural complications) | 11 | 13
Alanine aminotransferase increased (Investigations) | 15 | 17
Blood creatinine increased (Investigations) | 14 | 12
Anorexia (Metabolism and nutrition disorders) | 74 | 101
Dehydration (Metabolism and nutrition disorders) | 20 | 32
Hypokalaemia (Metabolism and nutrition disorders) | 13 | 10
Hyponatraemia (Metabolism and nutrition disorders) | 10 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 16
Dizziness (Nervous system disorders) | 38 | 34
Dysgeusia (Nervous system disorders) | 14 | 14
Headache (Nervous system disorders) | 46 | 48
Insomnia (Psychiatric disorders) | 14 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 15
Hiccups (Respiratory, thoracic and mediastinal disorders) | 63 | 74
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 16
Erythema (Skin and subcutaneous tissue disorders) | 13 | 4
Hypertension (Vascular disorders) | 17 | 6
Hypotension (Vascular disorders) | 11 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.